CLINICAL TRIAL: NCT06786988
Title: Cerebral Safety After Pulsed-Field Ablation of Atrial Fibrillation
Status: Not yet recruiting | Type: Observational
Sponsor: Charles University, Czech Republic (Other)
Responsible Party: Principal Investigator, Marek Hozman, MD, PhD, Interventional electrophysiologist, Charles University, Czech Republic
Other Study IDs: CNS_MRI_PFA
Record Dates: First submitted 2025-01-10; First posted 2025-01-22 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2025-01

CONDITIONS: Ischaemic Cerebral Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients undegoing AF ablation
  Interventions: Diagnostic Test: MRI

INTERVENTIONS:
Diagnostic Test: MRI — brain MRI scan: (1) one day before the procedure, (2) 24-36 hours after the procedure and (3) up to 1 year after the procedure

SUMMARY:
A study evaluating the incidence of ischaemic lesions detected by brain MRI scan in subjects undergoing pulsed-field ablation for atrial fibrillation (VARIPULSE system).

DETAILED DESCRIPTION:
An observational study evaluating the incidence of ischaemic lesions on brain MRI performed after ablation of atrial fibrillation using the Varipulse catheter.

1. A baseline MRI scan will be carried out one day before the procedure.
2. A post-procedure MRI scan will be performed 24-36 hours after the procedure.
3. A follow-up MRI will be performed within 1 year after the ablation.

Paroxysmal and non-paroxysmal AF patients will be included. Regarding the extent of ablation lesions, pulmonary vein isolation (PVI) will be performed in paroxysmal AF, whereas PVI + left atrial posterior wall ablation will be performed in non-paroxysmal patients. All procedures will be performed under intracardiac echocardiography guidance.

The patients will undergo a neurocognitive evaluation:

1. One day before the procedure: Montreal Cognitive Assessment (The MoCA Test)
2. 24-36 hours after the procedure: The National Institutes of Health Stroke Scale (NIHSS)
3. Up to 1 year after the procedure the MoCA test.

ELIGIBILITY:
Inclusion Criteria:

* AF with an indication for ablation

Exclusion Criteria:

* MRI contraindication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a common clinical indication for AF ablation.
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2025-02-01 (Estimated); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
ischaemic lesion | one day before the procedure (the first MRI scan), 24-36 hour sfter the procedure (the second scan) and up to 1 year after the procedure (the third scan)
  ischemic lesion on MRI

SECONDARY OUTCOMES:
Neurocognitive evaluation | one day before the procedure (the first MoCA test) and up to 1 year after the procedure (the second MoCA test)
  Change in the MoCA test result
NIHSS score | 24-36 hours after the procedure

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Laskov V, Hozman M, Malikova H, Lauer D, Kremenova K, Herman D, Hassouna S, Hornof J, Filipcova V, Vesela J, Waldauf P, Michalovova M, Karch J, Poviser L, Osmancik P. Cerebrovascular Ischemic Lesions After Pulsed Field Ablation for Atrial Fibrillation Using Variable-Loop Ablation Catheter. JACC Clin Electrophysiol. 2026 Jan 5:S2405-500X(25)01032-1. doi: 10.1016/j.jacep.2025.12.018. Online ahead of print. PMID 41575412